CLINICAL TRIAL: NCT06791278
Title: Improvements in Daily Activity and Exercise in School Children: the ActChild Study
Acronym: ActChild
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus Municipality, Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ActChild
Record Dates: First submitted 2024-12-17; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Healthy Children; Children; Children in School; Child Health; Child Behavior; Physical Activity; Sleep; Eating Behaviors; Child Obesity
Keywords: Exercise Intervention; Children; School Children; CEBQ; Eating Behavior; Sleep; Physical Activity; Quality of Life
MeSH Terms: conditions — Child Behavior; Motor Activity; Feeding Behavior; Pediatric Obesity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental study and participants will be assigned to intervention or control based on the time of inclusion. Each participating school will include controls at baseline. After one year, new participants will be included to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): 1-2 weekly sessions of 45-60 minutes of child-friendly exercise during after-school childcare programs. Duration: 1 year.
  Interventions: Behavioral: Exercise
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Exercise — After-school childcare educators will participate in a professional development course on delivering pedagogical and child-friendly exercise sessions. The children will receive 1-2 weekly sessions of 45-60 minutes of child-friendly exercise during after-school childcare programs. Duration: 1 year.
  Other Names: physical activity
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to assess the health-related effects of an exercise intervention in children aged 5-8 years.

Main research questions:

* Does a municipality-driven exercise intervention improve physical activity levels in children?
* Does a municipality-driven exercise intervention improve sleep parameters in children?
* Does a municipality-driven exercise intervention improve eating behaviors in children?
* Does a municipality-driven exercise intervention improve quality of life in children?

Study Design:

Participants will be assigned to either:

* Intervention group: Attend 1-2 weekly sessions of 45-60 minutes of child-friendly exercise for 1 year.
* Control group: Receive no intervention.

Data Collection:

Participants will:

* Complete questionnaires at baseline, and at 1-year, 3-year, and 5-year follow-ups.
* Wear accelerometers for 7 consecutive days at baseline, and at 1-year, 3-year, and 5-year follow-ups.

DETAILED DESCRIPTION:
Introduction:

Being physically inactive is associated with increased risk of developing non-communicable, lifestyle diseases such as Type 2 Diabetes (T2D), overweight/obesity, coronary heart disease (CHD) and premature death. In Denmark it is estimated that physical inactivity is responsible for more than 6000 deaths and related costs of 5.3 billion Danish Kroner each year. Although not fully elucidated, an increase in physical inactivity among children has over the last 20-30 years been observed in parallel with an increase in childhood overweight and obesity.

Aim:

The overall aim of this study is to promote (increase and sustain) healthy physical activity behaviors in children aged 5-8 years. The investigators wish to investigate the effects of an exercise intervention on physical activity, sleep (e.g. quality and duration), eating behavior, quality of life and anthropometrics.

Design The project is a collaborative clinical trial investigating the implementation of supervised physical activity in school children in Aarhus Municipality.

Intervention Children aged 5-8 years from Aarhus municipality will be included in the study. Initially first-year students from selected schools will be recruited as a control group. After one year an intervention group will be formed out of first-year students from the same schools. The intervention group will be invited to participate in a supervised training intervention during after-school daycare time.

The supervised physical activity will be conducted by after-school childcare educators in the municipalities, who have years of experience in handling children. The childcare educators will participate in a professional development course on delivering pedagogical and child-friendly exercise sessions.

Parents/legal guardians and participants will be able to withdraw from the study at any time.

Feasibility Feasibility and sustainability form the foundation of this exercise intervention. The project is developed, evaluated, and implemented in close collaboration with Aarhus Municipality. The intervention is designed to be easily maintained and scalable for implementation beyond the research setting.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren, 0.-1. Grade, 5-8 years of age,
* Resident in Aarhus Municipality

Exclusion Criteria:

- None

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-02-04 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Between group change in time spent in moderate to vigorous physical activity (MVPA) | Participants will wear accelerometers for 8 consecutive days at enrollment, and at 1-year, 3-year, and 5-year follow-ups
  Time spent in moderate to vigorous physical activity (MVPA). Physical activity levels will be measured with accelerometers (Axivity AX3) for 8 consecutive days. This will be repeated at each follow-up visit to compare changes in physical activity behavior between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of MVPA per day.
Between group change in total movement time | Participants will wear accelerometers for 8 consecutive days at enrollment, and at 1-year, 3-year, and 5-year follow-ups
  Total daily time the children spent moving in different body positions and engaging in different physical activities (standing, walking, running and biking). Physical activity levels will be measured with accelerometers (Axivity AX3) for 8 consecutive days. This will be repeated at each follow-up visit to compare changes in physical activity behavior between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of moderate to vigorous physical activity (MVPA) per day.
Between group change in time spent in light physical activity (LPA) | Participants will wear accelerometers for 8 consecutive days at enrollment, and at 1-year, 3-year, and 5-year follow-ups
  Time spent in light physical activity. Physical activity levels will be measured with accelerometers (Axivity AX3) for 8 consecutive days. This will be repeated at each follow-up visit to compare changes in physical activity behavior between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of moderate to vigorous physical activity (MVPA) per day.
Between group change in time spent being sedentary | Participants will wear accelerometers for 8 consecutive days at enrollment, and at 1-year, 3-year, and 5-year follow-ups
  Sedentary time is defined as any waking activity characterized as being in a sitting, reclining or lying posture with minimal stationary movement. Sedentary time will be measured with accelerometers (Axivity AX3) for 8 consecutive days. This will be repeated at each follow-up visit to compare changes in sedentary time between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of moderate to vigorous physical activity (MVPA) per day.
Between group change in total sleep time (TST) | Participants will wear accelerometers for 8 consecutive days at enrollment, and at 1-year, 3-year, and 5-year follow-ups
  Total sleep time will be measured with accelerometers (Axivity AX3) for 8 consecutive days. This will be repeated at each follow-up visit to compare changes in sleep parameters between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of moderate to vigorous physical activity (MVPA) per day.
Between group change in sleep efficiency (SE) | Participants will wear accelerometers for 8 consecutive days at enrollment, and at 1-year, 3-year, and 5-year follow-ups
  Sleep efficiency will be measured with accelerometers (Axivity AX3) for 8 consecutive days. This will be repeated at each follow-up visit to compare changes in sleep parameters between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of moderate to vigorous physical activity (MVPA) per day.
Between group change in sleep onset latency (SOL) | Participants will wear accelerometers for 8 consecutive days at enrollment, and at 1-year, 3-year, and 5-year follow-ups
  Sleep onset latency will be measured with accelerometers (Axivity AX3) for 8 consecutive days. This will be repeated at each follow-up visit to compare changes in sleep parameters between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of moderate to vigorous physical activity (MVPA) per day.
Between group change in wake after sleep onset (WASO) | Participants will wear accelerometers for 8 consecutive days at enrollment, and at 1-year, 3-year, and 5-year follow-ups
  Wake after sleep onset will be measured with accelerometers (Axivity AX3) for 8 consecutive days. This will be repeated at each follow-up visit to compare changes in sleep parameters between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of moderate to vigorous physical activity (MVPA) per day.

SECONDARY OUTCOMES:
Between group change in eating behavior | The CEBQ will be answered at enrollment, and at 1-year, 3-year, and 5-year follow-ups
  Eating behavior traits assessed by Children's Eating Behavior Questionnaire (the CEBQ). The CEBQ is a 35-item parent-report questionnaire assessing eating behavior in children. Eating behavior is assessed on eight scales: food responsiveness (4 items), enjoyment of food (4 items), emotional overeating (4 items), desire to drink (3 items), satiety responsiveness (5 items), slowness in eating (4 items), emotional undereating (4 items), and food fussiness (7 items). CEBQ responses will be scored from 1 to 5 and means for each subscale will be calculated. Changes in eating behavior will be compared between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of moderate to vigorous physical activity (MVPA) per day.
Between group changes in self-reported quality of life | Questionnaires will be answered at enrollment, and at 1-year, 3-year, and 5-year follow-ups.
  Quality of life will be assessed by the Pediatric Quality of Life Inventory (PedsQL). The PedsQL is a 23-item questionnaire with four Generic Core Scales: Physical Functioning (8 items), Emotional Functioning (5 items), Social Functioning (5 items) and School Functioning (5 items). Items on the PedsQL Generic Core Scales are reverse scored and transformed to a 0-100 scale. Higher scores indicate better health related quality of life. Two Summary Scores will be computed (the Psychosocial Health Summary Score and the Physical Health Summary Score), as well as a Total Scale Score. The Psychosocial Health Summary Score is the mean score on the Emotional, Social and School Functioning Scales. The Physical Health Summary Score is the mean score on the Physical Functioning Scale. The Total Scale Score is the mean of all items.
  A subsample analysis will be conducted on children who do not meet the WHO recommendations of 60 minutes of MVPA per day.
Between group change in BMI-SDS | From enrollment to the end of 5-year follow-up.
  Anthropometry data (i.e. heigth in cm, weight in kg and BMI in kg/m^2) measured from routine visits with the school health nurse will be transferred from Aarhus Municipality. Anthropometry data will be converted to standard deviation scores (BMI-SDS).
  Changes in BMI-SDS will be compared between intervention group and control group. A subsample analysis will be conducted on children who do not meet the WHO recommendation of 60 minutes of moderate to vigorous physical activity (MVPA) per day.
Baseline characteristics and data from school questionnaires | From enrollment to the end of the 5-year follow-up.
  Baseline characteristics is collected at enrollment. Aarhus Municipality will provide additional descriptive data from municipality-driven questionnaires (www.boernungeliv.dk).

CONTACTS AND LOCATIONS:
Overall Officials: Jens M Bruun, Professor, Principal Investigator — Aarhus University and Steno Diabetes Center Aarhus
Locations (1):
- Aarhus Municipality, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
The investigators have decided not to share individual participant data (IPD) due to ethical and privacy considerations, particularly given the sensitive nature of the data and the young age of the participants.